CLINICAL TRIAL: NCT05280418
Title: A Two-arm, Placebo-controlled, Randomized Clinical Trial to Evaluate the Effect of Tezepelumab on Airway Structure and Function in Patients With Uncontrolled Moderate-to-severe Asthma
Brief Title: Tezepelumab on Airway Structure and Function in Patients With Uncontrolled Moderate-to-severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-20-210000
Record Dates: First submitted 2022-02-11; First posted 2022-03-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Active Comparator): Tezepelumab 210 mg subcutaneous injections every 4 weeks as an investigational drug.
  Sterile tezepelumab will be provided 110 mg/mL pre-filled vial, with a dose of 210 mg delivered by pre-filled syringe.
  Interventions: Biological: Tezepelumab
- Matched placebo (Placebo Comparator): Sterile placebo for tezepelumab will be provided in identically matched pre-filled syringes.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Monoclonal antibody designed for the treatment asthma.
  Arms: Tezepelumab
Biological: Placebo — Matched placebo.
  Arms: Matched placebo

SUMMARY:
In adult patients with uncontrolled moderate-to-severe asthma, blocking TSLP with tezepelumab will improve ventilation heterogeneity (evaluated by hyperpolarized 129Xe MRI), and this will be associated with reduced airway inflammation (evaluated by sputum composition), luminal narrowing and plugging (evaluated by CT).

DETAILED DESCRIPTION:
The luminal obstruction in asthma that contributes to symptoms is due to inflammatory cells (usually eosinophils or neutrophils), mucus, smooth muscle constriction, airway wall thickness, or a combination of the above. This obstruction can be regionally visualized and quantified by computed tomography (CT), and its functional consequence can be assessed at high resolution using inhaled hyperpolarized 129Xe gas magnetic resonance imaging (MRI). Thymic stromal lymphopoietin (TSLP), an epithelial cell derived cytokine that is produced in response to environmental and proinflammatory stimuli, may contribute to all of these features of asthma through its downstream effects on a wide variety of immune (e.g. eosinophils, mast cells, group 2 innate lymphoid cells (ILC2s), Th2 cell, and Th17 cells) and structural cells (e.g. smooth muscle cells, and fibroblasts). Of note, TSLP is believed to upregulate multiple downstream inflammatory pathways, including IL-4, IL-5 and IL-13 signalling. It is also believed to mediate structural mechanisms that contribute to airway remodelling and smooth muscle dysfunction.

The consequence of blocking TSLP with tezepelumab on airway structure and function has not been investigated. This study will use CT to quantify airway wall and lumen structure according to previously described methods. CT images will also be evaluated for intraluminal plugging and a visual mucus score will be generated. Ventilation heterogeneity in asthmatics, the functional consequence of luminal obstruction, can be regionally measured with high temporal and spatial resolution using inhaled hyperpolarized gas MRI. In asthmatics, focal ventilation defects are observed and these have been shown to be spatially related to airway abnormalities and to respond to bronchoconstriction, bronchodilation, and anti-T2 biologics.

Due to the potential effect of tezepelumab on luminal inflammation, smooth muscle dysfunction and mucus hypersecretion, it is believed that MRI-detectable improvements in ventilation heterogeneity will be observed in asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* General

  * Able and willing to provide written informed consent.
  * Able and willing to comply with the study protocol.
  * Males and females ≥ 18 years of age.
* Asthma-related

  * Asthma diagnosed by a respiratory physician ≥12 months prior to study enrolment based on the Global Initiative for Asthma (GINA) 2021 guidelines.
  * ACQ ≥1.5 at screening.
  * Methacholine PC20 ≤ 4 mg/mL OR ≥15% decrease in FEV1 during saline inhalation for sputum induction OR ≥15% improvement in FEV1 after bronchodilator during the screening period.
  * Criteria met for moderate or severe asthma defined by GINA 2021 guidelines, i.e. treatment with low, medium or high dose ICS (<250 mcg, 251 - 500 mcg, >500 mcg of fluticasone equivalent/day respectively) plus another controller. Patients on prednisone would not be excluded, as long as they meet the rest of the inclusion criteria.
  * FeNO >25 ppb OR ≥3% sputum eosinophils (preferred) OR blood eos ≥300/µL during the screening period.
  * History of ≥1 exacerbation in the previous year.

Exclusion Criteria:

* General

  -- Participation in any clinical trial of an investigational agent or procedure within six months prior to screening or during the study.
* Medical conditions and treatment history

  * History of anaphylaxis to any previous biologic therapy received.
  * Receipt of live attenuated vaccine within 30 days, receipt of COVID vaccine within 28 days, known or suspected COVID infection at the time of enrollment.
  * Acute or chronic parasitic, bacterial, fungal or viral infections that required, or currently requires, hospitalization or antimicrobial treatment during the last four weeks.
  * Acute asthma exacerbation event treated with increased doses of oral, or any dose of intramuscular (IM) or intravenous (IV) corticosteroids within six weeks prior to screening.
  * Other relevant pulmonary diseases (e.g. chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis, pulmonary arterial hypertension, tuberculosis) requiring treatment within 12 months prior to screening.
  * Alcohol or substance abuse within 12 months prior to screening.
* Current smoker defined as having smoked at least one cigarette (or pipe, cigar, or marijuana) per day for ≥ 30 days within the three months prior to screening.

  * Ex-smokers with ≥ 10 pack-year smoking history.
  * Pregnancy.
  * Treatment with anti-IgE, anti-IL-4, anti-IL-5, or anti-IL-13 targeted therapy currently or within three months prior to screening.
* MRI-related

  * Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist).
  * In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Change in pre-bronchodilator 129Xe MRI ventilation defect percent (VDP). | 16 weeks from randomization (week 0) to endpoint assessment (week 16)
  Change from baseline to week 16 in the pre-bronchodilator 129Xe MRI ventilation defect percent (VDP).

SECONDARY OUTCOMES:
Change in the post-bronchodilator 129Xe MRI ventilation defect percent (VDP). | From baseline (week 0) to endpoint (week 16)
  Change in the post-bronchodilator 129Xe MRI ventilation defect percent (VDP) measured as percent of total ventilation.
Change in the CT mucus score (i.e. intraluminal plugging). | From baseline (week 0) to endpoint (week 16)
  Change in the CT mucus score (i.e. intraluminal plugging) measured using a mucus score.
Change in the CT airway lumen area. | From baseline (week 0) to endpoint (week 16)
  Change in the CT airway lumen area measured in mm^2.
Change in the CT airway wall area. | From baseline (week 0) to endpoint (week 16)
  Change in the CT airway wall area measured in mm^2.
Change in the CT airway wall area percentage. | From baseline (week 0) to endpoint (week 16)
  Change in the CT airway wall area percentage measured as a percentage of total airway area (wall area + airway lumen).
Change in the CT total airway count. | From baseline (week 0) to endpoint (week 16)
  Change in the CT total airway count
Change in the CT gas trapping. | From baseline (week 0) to endpoint (week 16)
  Change in the CT gas trapping
Change in the post-bronchodilator reversibility of 129Xe MRI VDP. | From baseline (week 0) to endpoint (week 16)
  Change in the post-bronchodilator reversibility of 129Xe MRI VDP measured by ventilation defect percentage of total ventilation

OTHER OUTCOMES:
Change in ACQ-5 score. | From baseline (week 0) to endpoint (week 16)
  Change in ACQ-5 score
Change in AQLQ score. | From baseline (week 0) to endpoint (week 16)
  Change in AQLQ score
Change in the pre-bronchodilator and post-bronchodilator FEV1. | From baseline (week 0) to endpoint (week 16)
  Change in the pre-bronchodilator and post-bronchodilator FEV1 measured in litres
Change in the post-bronchodilator reversibility of FEV1. | From baseline (week 0) to endpoint (week 16)
  Change in the post-bronchodilator reversibility of FEV1 measured in litres
Change in airways resistance and reactance measured by airwave oscillometry (R5, R20, R5-R20, X5, Ax). | From baseline (week 0) to endpoint (week 16)
  Change in airways resistance and reactance measured by airwave oscillometry (R5, R20, R5-R20, X5, Ax)
Change in FeNO. | From baseline (week 0) to endpoint (week 16)
  Change in FeNO measured as parts per billion
Change in blood eosinophil counts. | From baseline (week 0) to endpoint (week 16)
  Change in blood eosinophil measured as cells per litre
Change in blood neutrophil counts. | From baseline (week 0) to endpoint (week 16)
  Change in blood neutrophil counts measured as cells per litre
Change in sputum eosinophil counts. | From baseline (week 0) to endpoint (week 16)
  Change in sputum eosinophil counts measured as % total nucleated cells.
Change in sputum neutrophil counts. | From baseline (week 0) to endpoint (week 16)
  Change in sputum neutrophil counts measured as % total nucleated cells.
Change in eosinophil extracellular traps (including surrogate biomarkers histones, double stranded DNA and formalin fixed paraffin embedded sputum plugs). | From baseline (week 0) to endpoint (week 16)
  Change in absorbance values by fluorescence
Change in galectin-10 levels | From baseline (week 0) to endpoint (week 16)
  Change in galectin-10 concentration in sputum supernatant.
Change in sputum T2 cytokines. | From baseline (week 0) to endpoint (week 16)
  Change in sputum T2 cytokines.
Change in markers of airway eosinophil activity | From baseline (week 0) to endpoint (week 16)
  Change in eosinophil peroxidase (EPX) levels (ng/uL)
Change in markers of airway eosinophil activity | From baseline (week 0) to endpoint (week 16)
  Change in free eosinophil granules (FEGs) (none, few, moderate, many)

CONTACTS AND LOCATIONS:
Locations (1):
- Firestone Institute for Respiratory Health, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Gauvreau GM, Sehmi R, Ambrose CS, Griffiths JM. Thymic stromal lymphopoietin: its role and potential as a therapeutic target in asthma. Expert Opin Ther Targets. 2020 Aug;24(8):777-792. doi: 10.1080/14728222.2020.1783242. Epub 2020 Jun 27. PMID 32567399
- [Background] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- [Background] Svenningsen S, Haider E, Boylan C, Mukherjee M, Eddy RL, Capaldi DPI, Parraga G, Nair P. CT and Functional MRI to Evaluate Airway Mucus in Severe Asthma. Chest. 2019 Jun;155(6):1178-1189. doi: 10.1016/j.chest.2019.02.403. Epub 2019 Mar 23. PMID 30910637
- [Background] Menzies-Gow A, Corren J, Bourdin A, Chupp G, Israel E, Wechsler ME, Brightling CE, Griffiths JM, Hellqvist A, Bowen K, Kaur P, Almqvist G, Ponnarambil S, Colice G. Tezepelumab in Adults and Adolescents with Severe, Uncontrolled Asthma. N Engl J Med. 2021 May 13;384(19):1800-1809. doi: 10.1056/NEJMoa2034975. PMID 33979488